CLINICAL TRIAL: NCT06776731
Title: Hyperoxia During Outpatient Pulmonary Rehabilitation in Chronic Lung Disease - Does it Matter?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Switzerland University of Applied Sciences (Other)
Collaborators: University Hospital, Zürich (Other); Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: outRehaExO2
Record Dates: First submitted 2024-12-16; First posted 2025-01-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; oxygen therapy; pulmonary rehabilitation; hyperoxia; exercise medicine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Randomised, multicentre, double-blinded, sham-controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endurance training with 5l/ min room air applied via nasal cannula. (Placebo Comparator): Endurance training with 5l/ min room air applied via nasal cannula with an Everflo oxygen concentrator.
  Interventions: Other: Room Air (placebo)
- Endurance training with 5l/ min Oxygen Therapy applied via nasal cannula. (Experimental): Endurance training with 5l/ min Oxygen Therapy applied via nasal cannula with an Everflo oxygen concentrator..
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: Oxygen — Standard supplemental Oxygen therapy (5l/min) will be applied with an oxygen concentrator via nasal cannula during endurance training.
  Arms: Endurance training with 5l/ min Oxygen Therapy applied via nasal cannula.
Other: Room Air (placebo) — Room air (5l/min) will be applied with an oxygen concentrator via nasal cannula during endurance training.
  Arms: Endurance training with 5l/ min room air applied via nasal cannula.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a global burden. Treatment options have improved in recent years, pulmonary rehabilitation plays a key role. Oxygen therapy is recommended in patients with a low saturation at rest, but no clear guidance is given for patients who desaturate during exercise. The effect of ambulatory oxygen during exercise is not yet completely understood, especially in those patients with exercise-induced desaturation.

Aim: Evaluate the effect of supplemental oxygen therapy during a 3-months long ambulatory pulmonary rehabilitation program on exercise endurance. Patients will either receive supplemental oxygen therapy or room air during exercise training.

Methods: A total of 32 patients with a confirmed diagnosis of COPD undergoing pulmonary rehabilitation will be included (male and female : aged ≥ 18 years; stable condition > 3 weeks (e.g. no exacerbations); resting oxygen saturation (SpO2) ≥ 88% and exercise induced hypoxemia defined by a fall in SpO2 by ≥ 4% and/ or below 90% during a 6-minute walking test). 3-months comprehensive PR for both intervention and control group including: education and awareness, instruction on inhalation therapies, smoking cessation counselling, respiratory and skeletal muscle training in groups, guided walks / cycle ergometer training. The intervention group will be trained using SSOT and the control group will receive sham air (ambient air). Patients and assessors will be blinded. Between group difference in cycling constant work rate exercise test (CWRET) time from baseline to 3 months SSOT (5l/min) vs ambient air will be the primary outcome of this study.

Data will be summarized by means (SD) and medians (quartiles) for normal and non-normal distributions. Effects of treatment will be evaluated by mean differences with 95% confidence intervals, T-tests or Wilcoxon matched pair tests as appropriate. A p-value threshold of <0.05 or a confidence interval not including zero will be considered as statistically significant. Analyses will be performed according to the intention to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* We will include male and female with a confirmed diagnosis of COPD (post-bronchodilator forced expiratory volume in one second (FEV1) / forced vital capacity (FVC) ratio of <0.7; a greater than 10 pack-year smoking history)
* undergoing pulmonary rehabilitation
* aged ≥ 18 years
* stable condition > 3 weeks (e.g. no exacerbations)
* resting oxygen saturation (SpO2) ≥ 88%
* exercise induced hypoxemia defined by a fall in SpO2 by ≥ 4% and/ or below 90% during a 6MWT
* informed consent as documented by signature.

Exclusion Criteria:

* Severe daytime resting hypoxemia (SpO2 < 88% )
* long-term oxygen therapy, unstable condition requiring adaptation of pharmacologic and other treatment modalities or requirement of intensive care or relevant severe concomitant disease
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, neurological or orthopedic problems with walking disability or inability to ride a bicycle
* women who are pregnant or breast feeding; enrolment in another clinical trial with active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Constant Work Rate Exercise Test Endurance time | 3 months
  Constant Work Rate Exercise Test Endurance time measured with Constant Work Rate Exercise Test (CWRET) (75% of the maximal work rate from the maximal ramp exercise test)

SECONDARY OUTCOMES:
6 minute walk test (6MWT) | 3 months
  6 minute walk distance (6MWD), SpO2 and heart rate at the end of the 6 minute walk test (6MWT) from baseline to 3 months at SSOT vs ambient air
SpO2 | 3 months
  SpO2 by finger pulse oximetry, brain and muscle tissue oxygenation by NIRS at rest and end-exercise CWRET from baseline to 3 months at SSOT vs ambient air
Heart rate | 3 months
  Heart rate at rest and end-exercise CWRET from baseline to 3 months at SSOT vs ambient air
Borg scale | 3 months
  Borg scale (Dyspnoea and fatigue) at rest and end-exercise CWRET from baseline to 3 months at SSOT vs ambient air. Measure of perceived exertion from 1-10, ranges from 1 (very light exertion) to 10 (maximum exertion).
Constant Work Rate Exercise Test Endurance time | 6 months
  Constant Work Rate Exercise Test Endurance time measured with Constant Work Rate Exercise Test (CWRET) (75% of the maximal work rate from the maximal ramp exercise test)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof., Principal Investigator — University of Zurich
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request through the corresponding author